CLINICAL TRIAL: NCT01183975
Title: Prospective National Cohort Study on Swedish Adjustable Gastric Band (SAGB) for Gastroplasty (Étude de Cohorte Nationale Prospective de l'Implant Annulaire Ajustable Pour Gastroplastie SAGB)
Brief Title: Swedish Adjustable Gastric Banding Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-FR-004
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients treated with SAGB by solicited teams: Patients treated with SAGB by solicited teams. No selection criteria at cohort inclusion applied to the 500 (+50) first patients treated in order to ensure consecutive and exhaustive recruitment in the concerned centers over the inclusion period.

SUMMARY:
Longitudinal prospective cohort study of patients treated consecutively by SAGB in a sample of centers representative of this activity in France.

Verification by means of a screening log (exhaustive list of all bariatric procedures performed by participating surgeons between the beginning and end of the cohort inclusion period) requested from all centers.

No comparator group. No randomization or blinding techniques

DETAILED DESCRIPTION:
Longitudinal prospective cohort study of patients treated consecutively by SAGB in a sample of centers representative of this activity in France.

The study is originated in collaboration with HAS in France and has a target of 500 patients treated with gastric banding because of morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese patients (BMI>35 with comorbidities or BMI>40 without comorbidities) in France selected for gastric banding based on standard local clinical practice

Exclusion Criteria:

* lower BMI, contraindications based on local clinical assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is that of morbidly obese patients currently treated in France by gastroplasty (gastric banding with an SAGB). The CEPP notices define the indications in which this treatment is covered by health insurance.
Sampling Method: Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ribaric, MD,MSC,PhD, Study Director — Ethicon Endo-Surgery (Europe) GmbH
Locations (1):
- Polyclinique Rillieux, Rillieux-la-Pape, France

REFERENCES:
- [Derived] Ribaric G, Buchwald J. Gastric band is safe and effective at three years in a national study subgroup of non-morbidly obese patients. Croat Med J. 2014 Aug 28;55(4):405-15. doi: 10.3325/cmj.2014.55.405. PMID 25165055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The cohort consisted of 517 cases of the SAGB implanted by 31 surgeons recruited between 02 SEPT 2007 and 30 April 2008.
Period: Overall Study
Arm/Group | Patients Treated With SAGB by Solicited Teams
Started | 517
Completed | 444
Not Completed | 73
Not completed — Lost to Follow-up | 73

BASELINE CHARACTERISTICS:
Population: a longitudinal prospective cohort study of consecutive patients treated with SAGB in a representative sample of centers for this activity in France.
Arm/Group | Patients Treated With SAGB by Solicited Teams
Number analyzed (Participants) | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.92)
Gender [Number; unit: participants]
  Female | 455
  Male | 61
Region of Enrollment [Number; unit: participants]
  France | 517
Patients treated with SAGB by solicited teams [Number; unit: participants] | 517

OUTCOME MEASURES:

1. Primary Outcome: Mean BMI Change
Description: Mean change in BMI for valid subjects
Time Frame: 3 years follow-up
Population: 517 valid patients analyzed
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Patients Treated With SAGB by Solicited Teams
Number analyzed (Participants) | 517
kg/m^2 | -9.03 (5.31)

2. Primary Outcome: Mean Excess Weight Change
Description: Mean excess weight change in valid subjects. Excess weight is calculated as body weight minus ideal body weight, where ideal body weight is determined by the method of Lorentz (Ein neuer Konstitionsinde. Klin Wochenschr 1929; 8:348-51).
Time Frame: 3 years follow up
Measure: Mean (Standard Deviation); unit: percent change in excess weight
Arm/Group | Patients Treated With SAGB by Solicited Teams
Number analyzed (Participants) | 517
percent change in excess weight | -45.76 (29.97)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Patients Treated With SAGB by Solicited Teams
Serious Adverse Events (participants affected / at risk) | 123/517
Other Adverse Events (participants affected / at risk) | 26/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With SAGB by Solicited Teams (N=517)
Band Removal (Gastrointestinal disorders) | 67 (67) — Band Removal
abdominoplasty (Skin and subcutaneous tissue disorders) | 23 (23) — Abdominoplasty
port re-interventions without port removal (Gastrointestinal disorders) | 22 (22) — port re-interventions without port removal
port removal (Gastrointestinal disorders) | 8 (8) — Port Removal
band re-interventions without removal (Gastrointestinal disorders) | 3 (3) — band re-interventions without removal
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With SAGB by Solicited Teams (N=517)
band-related: Slippage (Gastrointestinal disorders) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less